CLINICAL TRIAL: NCT06624410
Title: Reduction of Perioperative Anxiety in Spanish-Speaking Children
Brief Title: We Will Compare Anxiety Levels Between English and Spanish-speaking Patients Before Surgery at a Children's Hospital. We Hypothesize That Spanish-speaking Patients Will Experience Greater Anxiety, so an Educational Intervention Will be Introduced One-week Before Surgery.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Tomas Lazo, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00024545; STUDY00024545 (Registry Identifier: eIRB)
Record Dates: First submitted 2024-09-23; First posted 2024-10-03 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-09

CONDITIONS: Anxiety; Healthcare Disparity
Keywords: anxiety; myPAS-SF; healthcare disparity
MeSH Terms: conditions — Anxiety Disorders | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Anesthesia providers, nurse providers, and surgical providers will be masked. The outcome assessor will be masked. The subject and their parent cannot be masked, due to the nature of the study. We will request of our subjects and parents/guardians to not inform their pre-operative nurse as to their allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): Pre-operative anxiety levels will be assessed with the mYPAS-SF6-12 (below). Subjects will be observed for behaviors and then given a score out of possible 5 across 5 domains that corresponds with demonstrated behaviors, specified in the figure below. The 5 domains include Activity, Vocalization, Emotional Expressivity, State of Arousal, and Use of Parent. Note that the "Vocalization" domain differs in that It's possible scores range from 1-7. Pilot data collection will involve mYPAS scoring in isolation to demonstrate existing anxiety burden at Doernbecher Children's Hospital.
- Educational Intervention Arm (Experimental): The educational intervention, an informational video to prepare the child for what to expect in the perioperative period, will be delivered within one week of the scheduled surgery assuming parental consent has been confirmed. They will watch the video prior to coming in for surgery and then proceed to have standard care provided as they are assessed for anxiety scores.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Pre-operative anxiety levels will be assessed with the mYPAS-SF6-12 (below). Subjects will be observed for behaviors and then given a score out of possible 5 across 5 domains that corresponds with demonstrated behaviors, specified in the figure below. The 5 domains include Activity, Vocalization, Emotional Expressivity, State of Arousal, and Use of Parent. Note that the "Vocalization" domain differs in that It's possible scores range from 1-7. Pilot data collection will involve mYPAS scoring in isolation to demonstrate existing anxiety burden at Doernbecher Children's Hospital.
  Arms: Educational Intervention Arm

SUMMARY:
The goal of this trial is to first evaluate whether a difference exists in anxiety scores between Spanish-speaking children and English-speaking children in the pre-operative setting in our patient population as assessed by the validated myPAS-SF anxiety index. In the interventional phase, the investigators hypothesize that the use of a language-concordant, educational intervention by study participants at home during the week preceding surgery will decrease pre-operative anxiety in Spanish-speaking children, as assessed by the validated mYPAS-SF anxiety index.

DETAILED DESCRIPTION:
Rationale: Pre-operative anxiety is a common phenomenon among children as well as their parents with some studies suggesting it occurs in up to 50% of children who are undergoing surgery in the United States (U.S.). Therefore, the prevalence of this phenomenon within the surgical field represents a solvable problem, the elimination of which would be of added benefit to the surgical experience for patients. Beyond the simple unpleasantness of experiencing anxiety, higher levels of pre-operative anxiety have also been shown to associate with worse post-surgical outcomes including increased pain, agitated emergence from anesthesia (emergence delirium) and maladaptive behavioral change. Indeed, this means that addressing pre-operative anxiety could lead to better overall health outcomes post-operatively.

Demographically, the Hispanic / Latino population is one of the fastest growing in the U.S., with a predicted increase by 240% by the year 2060, meaning that one in three US residents will be Hispanic at that time. Our ever-diversifying US population highlights a need for more personalized and culturally considerate medical care, as research has shown that ethnicity, culture, and language may play a role in decision making as well as the patient experience.

Given the association between pre-operative anxiety and worse post-operative outcomes and the fact that Hispanic children with Spanish-speaking parents experience higher levels of pre-operative anxiety as opposed to their white counterparts, the investigators have thus identified a gap in healthcare that leaves Hispanic populations vulnerable to preventable health disparities. Therefore, the purpose of this project is to create an intervention designed specifically for Hispanic, Spanish-speaking children that will lower rates of pre-operative anxiety and thus improve their post-operative outcomes.

Background: To address the problem of pre-operative anxiety in children, it was paramount to develop a valid metric for accurately assessing anxiety level. To assist with measuring anxiety in children before surgery, the modified Yale Preoperative Anxiety Scale (mYPAS) was developed in 1995 and then modified in 1997. This scale uses 5 items, each of which represent a different domain of child anxiety and is used at 4 distinct timepoints throughout the surgical experience. However, though this metric was reliable and accurate, the inclusion of 5 different domains of assessment over 4 timepoints proved to be somewhat redundant and cumbersome to use in a hectic surgical setting. Therefore, in 2014, Jenkins et al. developed a short form version of the mYPAS, aptly renamed mYPAS-SF through elimination of areas of redundancy and only administered at 2 time points instead of 4. Use of this metric has helped identify characteristics which may correspond to higher levels of anxiety such as younger age, a shyer temperament, an established history of surgery, and miscellaneous parental factors.

Once a reliable metric for assessing pre-operative anxiety in children was established, various experimental interventions were developed and introduced to children pre-operatively like listening to calming music or encouragement of participation in recreation beforehand, both of which had a significant impact on the reduction of pre-operative anxiety. However, an inherent problem with these studies is that most of them are conducted on primarily white, English-speaking children or their parents which limits their generalizability. Indeed, research has confirmed that cultural consideration is necessary; Hispanic children with Spanish-speaking parents experience higher levels of pre-operative anxiety as compared to white children with English-speaking parents. This is not exclusively limited to children, but to their parents as well. Fortier et al., specifically concluded that "Spanish-speaking Hispanic parents exhibited higher levels of anxiety and this correlates to higher levels of preoperative anxiety in their children". These differences represent a gap in healthcare that could be filled through tailored delivery of interventions pre-operatively which reduce Hispanic children's anxiety and will correspond to better outcomes post-operatively.

Study Design: Initially, the investigators plan to perform an observational pilot study to identify differences in pre-operative anxiety scores in our patient population between English-speaking patients and Spanish-speaking patients. This will not include any sort of intervention, only generation of mYPAS scores between two groups of patients. The investigators will use the same inclusion and exclusion criteria for this phase, with the goal of identifying 20 patients in each arm.

The main study to follow our pilot data gathering phase is a single center, prospective, randomized controlled trial (RCT) with 1:1 allocation between 2 parallel arms. Blocked randomization will be used to reduce bias, reduce the opportunity for confounding, and achieve balance between study arms. To reduce selection bias, random block sizes of 4 and 8 will be used, with blinding of the investigator to block size.

Intervention arm: Home video educational intervention Control arm: Standard of care preoperative instructions

The initial observational phase of the study will look at 20 English-speaking children in comparison with 20 Spanish-speaking children and their mYPAS scores. This will be to help elucidate any existing difference in baseline anxiety between groups. Investigators will then move onto the intervention portion of the study by implementing an educational home video for Spanish-speaking families to watch in preparation for the surgery.

For both the observational and intervention portion of the study, baseline anxiety will be scored by the mYPAS scoring system, with a range of 23-100 as an anxiety score. Prior studies noted that a score in the 40s is predictive for worsened anxiety at induction of anesthesia, where a score of >60 was associated with extreme anxiety. Thus, a decrease in anxiety score of 10-15 may be argued as valuable. From prior studies, investigators have noted about a 30% decrease with their interventions. Based on pilot data collected from our DCH patient population, investigators have decided on the numbers below to find a similar difference based on power analysis calculations. The portion of the study will include 25 subjects in the intervention arm and 25 subjects in the control (standard of care) arm. Investigators will aim to enroll more patients to improve our sample size as able from the Doernbecher hospital on the OHSU campus. The investigators predict that 5-10% of patients within the Doernbecher operating room will meet inclusion criteria and assume a 50% enrollment rate to achieve a total enrollment number of around 50 patients.

Strategies for Subject Recruitment and Retention: Most subject recruitment is expected to occur by approved study staff the week prior to surgery in Doernbecher Children's Hospital via review of the surgical schedule as posted in Epic (Verona, Wisconsin). The investigators will work with anesthesiology providers and pre-anesthesia nursing staff to identify and screen for potential eligible subjects. All inclusion/exclusion criteria will be reviewed as early as two weeks prior to a potential subject's scheduled surgery. If a potential subject has been identified as meeting all inclusion criteria and none of the exclusion criteria, an approved member of the study team will call the potential subject's parent using the approved telephone script to introduce the study (included in 'Consent Form and Recruitment Materials' section of application). If the subject's parent is amenable to including the subject in the study, study staff will provide formal consent materials and obtain signature. Spanish-speaking subjects will be consented and enrolled using phone interpretive services.

Vulnerable Populations: The clinical question is about children, so it is impossible to conduct this study without involving children. Vulnerable populations including neonates (up to 28 days post birth) will be excluded. Children currently in youth correctional facilities and pregnant pediatric subjects in our age range will be excluded.

Setting: The study will take place in the pediatric operating suites of OHSU (Doernbecher Hospital), located in Portland, Oregon. Verbal consent will be obtained through the telephone during the week preceding surgery. All study interventions will occur in the preoperative area, the operating rooms, or in the post-anesthesia care unit. Data collection will continue to occur throughout the patient's hospitalization.

Consent Process: The subject parent consent process will take place over the phone with the research staff in a private and confidential area. All subject parents that are approached for recruitment will hear a description of the study, reasons for pursuing this research study, options for opting out the research protocol or not completing data collection, and potential risks, advantages, and disadvantages from participating. Investigators will ask pediatric subjects to reiterate their understanding of how the study will affect their care and allow time for questions. If subject age and mental capacity allow, assent will be obtained from study subjects. A copy of the consent will be mailed electronically to subjects for their medical records.

Since this study poses no more than minimal risk and no procedures will be conducted in this study, for which written documentation is normally required, outside of research, verbal consent will be used in lieu of written consent. Due to the minimal risk nature of the study, permission from one parent or guardian will be sufficient. The study team will identify parents who are able to assent based on age and cognitive ability and present all necessary consent information and documentation to them. Both parental consent and subject assent will be documented in the HIPAA compliant database. After verbal consent has been obtained an informational sheet will be emailed to subject parents. The informational sheet will be created in both Spanish and English.

Investigators are requesting that verbal consent be used for this study because it is not practical to obtain consent prior to the day of surgery. Verbal consent will not adversely affect the rights or welfare of the study subjects. Investigators will provide contact information for the principal investigator on the informational sheet and study subjects, and their parents, will be informed on how to withdrawal, without penalty, from the study at any time.

For study subjects, or their parents, who are not primary English speakers, consent documentation will be communicated verbally over the phone in the subject's native language, with 3rd party medical grade interpretation or a certified interpreter from the study team. Interpreter services will be used for all study visits.

Handling of Data: Study subjects will be assigned a unique study number after enrollment in the study. All data points, procedure related data, and electronic files for data analysis will be linked only to this unique study number which will be not include patient identifying information. The key linking study subjects to study code will be kept in a cloud location with special protection for confidential and restricted health information (the OHSU OneDrive) for indefinite use. Only the principal investigator and other study staff will have access to this key.

Data Analysis: The database will be created and managed by Praveen Tekkali, a computer scientist within the Clinical Research Division of Anesthesiology and Perioperative Medicine. The statistical analysis described herein will be conducted by RDB. The research team led by Dr. Tomas Lazo will be responsible for interpreting the data.

Statistical Analysis: The primary endpoints of this study will be pediatric patient preoperative anxiety, measured in the pre-operative bay while awaiting surgery, with the mYPAS-SF anxiety index. Simple descriptive statistics and the student T-test or Mann Whitney test will be used where appropriate. All statistical analysis will use intention-to-treat patient population.

Power/Sample Size: This study is powered to detect a 30% percent reduction in preoperative anxiety, as measured by the mYPAS-SF anxiety index. Our baseline mYPAS-SF anxiety for pediatric patients at Doernbecher is 38.6. As such, investigators plan to enroll 25 subjects in each arm.

Privacy, Confidentiality and Data Security: Verbal consent will be obtained from parents interested in participating over the phone. The research team will conduct these phone interviews from closed private offices in Multnomah Pavilion, 3rd floor. Phone calls be made from OHSU phones using approved OHSU long distance codes. The key linking study subjects to study code will be kept in a cloud location with special protection for confidential and restricted health information (OHSU OneDrive). Only the principal investigator and other study staff will have access to this key.

Potential Benefits to Subjects: This study is being performed because preoperative anxiety has been linked to worse postoperative outcomes and pediatric non-English speakers have higher levels of preoperative anxiety. Patients in the intervention group may experience lower preoperative anxiety and have greater understanding of perioperative anesthesia care.

Risks and Benefits Risks to Subjects: As with all studies, breach of confidentiality is a common risk. In addition, there is the possibility of slightly increased anxiety or psychological stress on the day of surgery. Investigators believe the magnitude and duration of this psychological stress to be small and brief. There is also likely to be a loss of free time in the preoperative area due to study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic/Latino Spanish-Speaking children ages 5-14 years
* Undergoing surgery in the Doernbecher Operating Rooms

Exclusion Criteria:

* Subjects having cardiac surgery
* Parent refusal of consent
* Children that refuse assent
* Children with psychiatric or atypical neurodevelopmental conditions such as autism or sensory processing disorders that put them at greater risk for pre-surgical anxiety, history of prior surgery, and children with global developmental delay as noted by ICD codes or diagnosis on their problem list

Parent/Guardian Exclusion Criteria

* Impaired decision-making adults
* Incarcerated adults

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety score using the mYPAS-SF anxiety index | On average 1-2 weeks. From enrollment to day of surgery.
  Pre-operative anxiety levels will be assessed with the mYPAS-SF6-12 (below). Subjects will be observed for behaviors and then given a score out of possible 5 across 5 domains that corresponds with demonstrated behaviors, specified in the figure below. The 5 domains include Activity, Vocalization, Emotional Expressivity, State of Arousal, and Use of Parent. Note that the "Vocalization" domain differs in that It's possible scores range from 1-7. Pilot data collection will involve mYPAS scoring in isolation to demonstrate existing anxiety burden at Doernbecher Children's Hospital.

SECONDARY OUTCOMES:
Post-operative/Emergence Delirium | Up to 24 hours
  Defined as an altered state of consciousness, which begins with emergence from anesthesia and continues through the early recovery period. ED is a disturbance of awareness of, or attention to, the child's environment, and manifests as disorientation, hyperactive behavior, and hypersensitivity in the immediate period after anesthesia.
VAS pain score | Up to 1 week
  Initial visual analog pain score recorded by the recovery room nurse
Morphine equivalents | Up to 1 week
  Parental morphine equivalents administered during phase I of the post-anesthesia care unit-these have all been associated with anxiety

OTHER OUTCOMES:
PACU phase 1 duration | From day of surgery to end of recovery period in the post-anesthesia care unit
  Time spent in phase 1 in the recovery area
Total PACU duration | Up to 1 week.
  Total time spent in the recovery unit, including phase 1 and phase 2 of recovery

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Togioka, MD, Study Chair — Oregon Health & Science University

IPD SHARING:
Plan to Share IPD: No
Plan to keep data centralized and kept within our hospital and department. We do not plan to share data at this time.

REFERENCES:
- [Background] Mamtora PH, Kain ZN, Stevenson RS, Golianu B, Zuk J, Gold JI, Fortier MA. An evaluation of preoperative anxiety in Spanish-speaking and Latino children in the United States. Paediatr Anaesth. 2018 Aug;28(8):719-725. doi: 10.1111/pan.13425. Epub 2018 Jul 1. PMID 29962037
- [Background] Fortier MA, Gomez SH, Kain A. Motivation and parental presence during induction of anesthesia: an examination of the role of ethnicity and language. Paediatr Anaesth. 2012 Nov;22(11):1094-9. doi: 10.1111/j.1460-9592.2012.03841.x. PMID 22458854
- [Background] Weber FS. The influence of playful activities on children's anxiety during the preoperative period at the outpatient surgical center. J Pediatr (Rio J). 2010 May-Jun;86(3):209-14. doi: 10.2223/JPED.2000. Epub 2010 Apr 23. PMID 20419272
- [Background] Franzoi MA, Goulart CB, Lara EO, Martins G. Music listening for anxiety relief in children in the preoperative period: a randomized clinical trial. Rev Lat Am Enfermagem. 2016 Dec 19;24:e2841. doi: 10.1590/1518-8345.1121.2841. PMID 27992027
- [Background] Vetter TR. The epidemiology and selective identification of children at risk for preoperative anxiety reactions. Anesth Analg. 1993 Jul;77(1):96-9. doi: 10.1213/00000539-199307000-00019. PMID 8317755
- [Background] Kain ZN, Mayes LC, Weisman SJ, Hofstadter MB. Social adaptability, cognitive abilities, and other predictors for children's reactions to surgery. J Clin Anesth. 2000 Nov;12(7):549-54. doi: 10.1016/s0952-8180(00)00214-2. PMID 11137417
- [Background] McCann ME, Kain ZN. The management of preoperative anxiety in children: an update. Anesth Analg. 2001 Jul;93(1):98-105. doi: 10.1097/00000539-200107000-00022. No abstract available. PMID 11429348
- [Background] Fortier MA, Del Rosario AM, Martin SR, Kain ZN. Perioperative anxiety in children. Paediatr Anaesth. 2010 Apr;20(4):318-22. doi: 10.1111/j.1460-9592.2010.03263.x. Epub 2010 Feb 23. PMID 20199609
- [Background] Jenkins BN, Fortier MA, Kaplan SH, Mayes LC, Kain ZN. Development of a short version of the modified Yale Preoperative Anxiety Scale. Anesth Analg. 2014 Sep;119(3):643-650. doi: 10.1213/ANE.0000000000000350. PMID 25010821
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Kain ZN, Caldwell-Andrews AA, Mayes LC, Weinberg ME, Wang SM, MacLaren JE, Blount RL. Family-centered preparation for surgery improves perioperative outcomes in children: a randomized controlled trial. Anesthesiology. 2007 Jan;106(1):65-74. doi: 10.1097/00000542-200701000-00013. PMID 17197846
- [Background] Perry JN, Hooper VD, Masiongale J. Reduction of preoperative anxiety in pediatric surgery patients using age-appropriate teaching interventions. J Perianesth Nurs. 2012 Apr;27(2):69-81. doi: 10.1016/j.jopan.2012.01.003. PMID 22443919
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995